CLINICAL TRIAL: NCT04703647
Title: Longitudinal Follow-up Study About Complex Regional Pain Syndrome (CRPS). Which Are the Predictors for Return to Work and Recovery
Brief Title: Longitudinal Follow-up Study About Complex Regional Pain Syndrome (CRPS) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Other Study IDs: CliniqueRR-20
Record Dates: First submitted 2020-12-09; First posted 2021-01-11 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-08

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: pain; biopsychosocial model; miRNAs; cytokines; upper limb; lower limb
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain | interventions — Blood Specimen Collection; Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For patients, blood samples will be collected at T0 (beginning of the study), T1 (3 months after T0) and, T2 (6 months after T0) and T3 (1 year after T0) by the study nurse (each time two 7.5 ml S-Monovette® K3 EDTA tubes).The samples will be first coded and then processed in our laboratory. After processing, samples will be stored at -80°C in a secured freezer. MiRNAs and various cytokines will be measured directly in our laboratory in Sion using previous validated protocols.
  For controls (30 patients) will be collected blood samples just one time for comparison with the patients. These same analysis than patients will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CRPS type 1: prospective group: Ambulatory patients of the Clinique romande de réadaptation (CRR) which have a CRPS type 1 of a limb.
  Five measurement times (first visit (T0) and then after 3 (T1), 6 (T2), 12 (T3) and 24 (T4) months). At every time point, following data will be collected: physical examination, monitoring of the health and professional status with the physician, and self-administrated questionnaires. Blood sampling will be performed at T0, T1,T2 and T3.
  Eight different self-administrated questionnaires will be used, in their French or Portuguese version. Each participants will answer seven questionnaires each time, depending if he/she suffers of arm or leg injury.
  We will assess, in blood samples, the expression levels of specific molecules (miRNAs and a selection of cytokines) in patients diagnosed with acute CRPS. In a second time, miRNAs and cytokines profiles will be compared between acute and chronic (CRPS still diagnosed 6 months after the first diagnosis) CRPS patients.
  Interventions: Other: Administration of questionnaires for prospective group; Other: Blood samples for prospective group
- control group for blood analysis: For the blood analysis, we will recruit 30 healthy controls who did not report any kind of pain. They will be recruited via posters that will be posted on the billboards of the Hôpital de Sion (employees and visitors) and on the visitor's billboards of the CRR. If this is not enough, we will expand the recruitment perimeter with other locations. The healthy control will be adjusted for age, sex and BMI with the CRPS groups. They will be informed about the study and procedure. The procedure for the blood samples will be the same as for patients.The screening for miRNAs of interest will be performed using a decision tree-based ensemble method (Random Forest). For this step, miRNAs profile of 30 control patients will be compared to the same number of CRPS patients.
  The control group will have just one blood analysis.
  Interventions: Other: Blood samples for control group

INTERVENTIONS:
Other: Administration of questionnaires for prospective group — Questionnaires: administration at T0, T1,T2,T3 and T4 of Short Form Health Survey (SF-36),Brief Pain Inventory (BPI),Disabilities of the Arm, Shoulder and Hand (DASH) for upper limb,Foot and Ankle Ability Measure (FAAM) for lower limb,Hospital Anxiety And Depression Scale (HADS),Tampa Scale of Kinesiophobia (TSK),Pain Catastrophizing Scale (PCS),Pattern Of Activity Measure - Pain (POAM-P) .
  Groups: Patients with CRPS type 1: prospective group
Other: Blood samples for prospective group — Blood samples at T0,T1,T2 and T3.
  Groups: Patients with CRPS type 1: prospective group
Other: Blood samples for control group — Blood samples just one time
  Groups: control group for blood analysis

SUMMARY:
Complex regional pain syndrome (CRPS) is a post-traumatic chronic pain condition characterized by pain and other symptoms typically affecting a distal limb. Relatively little is known about the prognosis of the course of CRPS .Currently there is no specific test to diagnose CRPS.

The primary objective of the study is to investigate prospectively the evolution of CRPS and the impact of the psychosocial factors on health status, recovery, quality of life, and working status of CRPS patients.

The secondary objective of the study is to measure blood parameters in CRPS patients to investigate their evolution during the course of CRPS, and maybe to identify distinctive biomarkers associate with CRPS and that could be potential candidate for diagnosis.

DETAILED DESCRIPTION:
The first aim will be to monitor the evolution of the following parameters in CRPS patients:

* Quality of life
* Symptoms and signs of CRPS
* Severity of CRPS
* Working status
* Pain
* Disability
* Anxiety and depression
* Kinesiophobia
* Catastrophism
* Activity patterns with chronic pain during the two years follow-up. Every parameter will be evaluated with a questionnaire that allows assigning scores to each patient.

Additionally sociodemographic data will be collected to characterize the patients (age, gender, marital status, educational level). The health status, treatment and medication of the patients will also be recorded with a medical follow-up during the two years.

The aim is to know if the following parameters and their evolution:

* Sociodemographic factors,
* Pain,
* Disability,
* Anxiety and depression,
* Kinesiophobia,
* Catastrophism,
* Activity patterns with chronic pain

are associated with the recovery, which is evaluated with

* Quality of life,
* Severity of CRPS,
* And working status.

Potential associations between the different parameters will be tested (Pearson's correlation coefficient).

The second aim will be to assess, in blood samples, the expression levels of specific molecules (miRNAs and a selection of cytokines) in patients diagnosed with acute CRPS. Comparison with healthy controls will be performed at the first measurement time (T0) . In a second time, miRNAs and cytokines profiles will be compared between acute and chronic (CRPS still diagnosed 6 months after the first diagnosis) CRPS patients. The measured proteins will include: C-reactive protein, tumor necrosis factor-alpha (TNF), interleukin-2 [IL-2], IL-6, IL-8, IL-10, CD40 ligand (pro- and anti-inflammatory proteins associated with pain), gene related peptide (CGRP), bradykinins and substance P.

The screening, recruitment and enrolment of the patients will be done by the referring physician in daily clinical practice, during the consultation.

The physician will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail. Each participant will be informed that the participation in the study is voluntary and that he/she may withdraw from the study at any time and that withdrawal of consent will not affect his/her subsequent medical assistance and treatment.

All participants for the study will be provided with a participant information sheet,a consent form describing the study and providing sufficient information for participant to make an informed decision about their participation in the study and a prepaid envelope. Each patient may decide separately to participate in a) longitudinal follow-up questionnaires, b) blood tests or c) both parts of the study (questionnaire and blood samples). The delay for reflection will be 24 h. Once this period has expired, if the patient agrees to participate in the study, he or she is asked to return the consent form in the prepaid envelope. If he or she has not been send back after one week, the physician will call the patient by phone to make sure that it is not an omission.

The patient information sheet and the consent form are submitted to the Ethic comitee to be reviewed and approved. The formal consent of a participant, using the approved consent form, must be obtained before the participant is submitted to any study procedure.

The participant should read and consider the statement before signing and dating the informed consent form, and should be given a copy of the signed document. If the patient sent back the informed consent, a next appointment will be scheduled at the CRR where he or she will be asked to submit the signed consent form. The consent form must also be signed and dated by the investigator (or his designee) and it will be retained as part of the study records.

The total duration of the project is planned over a six years period (2019-2024). The study will be proposed to every CRPS ambulatory patient in the CRR (2019-2022), inclusion period). The study will also be proposed to the patients during the last two years (2023-2024) but only partially, since that last questionnaires will be sent in December 2024.

The CRPS patients are monitored on a regular and long-term basis at the CRR. The physician see them very regularly at the beginning (about once a month) and then the visits space a little out. Thus, our study fits into routine procedure and should not imply additional visits.

At the first visit at the clinic, the physician will proposed the study to the patient. Upon acceptance, the patient will be included into the study. It consists in five measurement times:

* T0: During the days following the first visit to the clinic
* T1: Follow up visit 3 months later
* T2: Follow up visit 6 months later
* T3: Follow up visit 12 months later
* T4: Follow up visit 24 months later

ELIGIBILITY:
Inclusion Criteria for patients:

* CRPS Type I (fulfilling Budapest criteria for research)
* Suffering of CRPS in a distal limb (hand or foot)
* Age >18 years
* Pain lasting less than 6 months
* Good understanding of the French language

Inclusion criteria for control:

* Not suffering from chronic pain, including CRPS
* Age >18 years

Exclusion Criteria for both group:

* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, severe psychological disorders, dementia, etc
* For blood sample: diabetes and history of hepatitis B, C, D or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited among the patients admitted for acute CRPS of the upper or lower limb in the CRR. It will be only ambulatory patients.The screening, recruitment and enrolment of the patients will be done by the referring physician in daily clinical practice, during the consultation.
  For control group (blood analysis) we will recruit 30 healthy controls who did not report any kind of pain. The healthy control will be adjusted for age, sex and BMI with the CRPS groups. They will be informed about the study and procedure. The procedure for the blood samples will be the same as for patients.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
patient return to work (RTW) | 3 months after inclusion
  Percentage of patients return to work at T1
patient return to work (RTW) | 6 months after inclusion
  Percentage of patients return to work at T2
patient return to work (RTW) | 1 year after inclusion
  Percentage of patients return to work at T3
patient return to work (RTW) | 2 years after inclusion
  Percentage of patients return to work at T4
Recovery of CRPS | 3 months after inclusion
  Disability of the patients evaluated with DASH questionnaire for upper limb and FAMM questionnaire for lower limb at T1. For DASH the score range from 0 to 100, with 100 represent the worst disability. For FAMM the score range from 0 to 100, 100 represent the best functionality.
Recovery of CRPS | 6 months after inclusion
  Disability of the patients evaluated with DASH questionnaire for upper limb and FAMM questionnaire for lower limb at T2. For DASH the score range from 0 to 100, with 100 represent the worst disability. For FAMM the score range from 0 to 100, 100 represent the best functionality.
Recovery of CRPS | 1 year after inclusion
  Disability of the patients evaluated with DASH questionnaire for upper limb and FAMM questionnaire for lower limb at T3. For DASH the score range from 0 to 100, with 100 represent the worst disability. For FAMM the score range from 0 to 100, 100 represent the best functionality.
Recovery of CRPS | 2 years after inclusion
  Disability of the patients evaluated with DASH questionnaire for upper limb and FAMM questionnaire for lower limb at T4. For DASH the score range from 0 to 100, with 100 represent the worst disability. For FAMM the score range from 0 to 100, 100 represent the best functionality.

SECONDARY OUTCOMES:
miRNAs and cytokines profile of patients and control | at T0 (after inclusion)
  Mesure in blood samples of miRNAs and cytokines in patients and 30 healthy control at T0
miRNAs and cytokines profile of patients | 3 months after inclusion
  Mesure in blood samples of miRNAs and cytokines in patients at T1
miRNAs and cytokines profile of patients | 6 months after inclusion
  Mesure in blood samples of miRNAs and cytokines in patients at T2
miRNAs and cytokines profile of patients | 1 year after inclusion
  Mesure in blood samples of miRNAs and cytokines in patients at T3

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Léger, PhD, Study Director — institut de recherche en réadaptatation
Locations (1):
- Clinique romande de réadaptation, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Protocol of the study

REFERENCES:
- [Background] Konig S, Schlereth T, Birklein F. Molecular signature of complex regional pain syndrome (CRPS) and its analysis. Expert Rev Proteomics. 2017 Oct;14(10):857-867. doi: 10.1080/14789450.2017.1366859. Epub 2017 Aug 17. PMID 28803495
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633
- [Background] Orlova IA, Alexander GM, Qureshi RA, Sacan A, Graziano A, Barrett JE, Schwartzman RJ, Ajit SK. MicroRNA modulation in complex regional pain syndrome. J Transl Med. 2011 Nov 10;9:195. doi: 10.1186/1479-5876-9-195. PMID 22074333
- [Background] Galer BS, Henderson J, Perander J, Jensen MP. Course of symptoms and quality of life measurement in Complex Regional Pain Syndrome: a pilot survey. J Pain Symptom Manage. 2000 Oct;20(4):286-92. doi: 10.1016/s0885-3924(00)00183-4. PMID 11027911
- [Background] Bean DJ, Johnson MH, Heiss-Dunlop W, Kydd RR. Extent of recovery in the first 12 months of complex regional pain syndrome type-1: A prospective study. Eur J Pain. 2016 Jul;20(6):884-94. doi: 10.1002/ejp.813. Epub 2015 Nov 2. PMID 26524108
- [Background] Bean DJ, Johnson MH, Heiss-Dunlop W, Kydd RR. Factors Associated With Disability and Sick Leave in Early Complex Regional Pain Syndrome Type-1. Clin J Pain. 2016 Feb;32(2):130-8. doi: 10.1097/AJP.0000000000000234. PMID 25803756
- [Background] Bean DJ, Johnson MH, Heiss-Dunlop W, Lee AC, Kydd RR. Do psychological factors influence recovery from complex regional pain syndrome type 1? A prospective study. Pain. 2015 Nov;156(11):2310-2318. doi: 10.1097/j.pain.0000000000000282. PMID 26133727
- [Background] Birklein F, Ajit SK, Goebel A, Perez RSGM, Sommer C. Complex regional pain syndrome - phenotypic characteristics and potential biomarkers. Nat Rev Neurol. 2018 May;14(5):272-284. doi: 10.1038/nrneurol.2018.20. Epub 2018 Mar 16. PMID 29545626
- [Background] Le Carre J, Lamon S, Leger B. Validation of a multiplex reverse transcription and pre-amplification method using TaqMan((R)) MicroRNA assays. Front Genet. 2014 Nov 26;5:413. doi: 10.3389/fgene.2014.00413. eCollection 2014. PMID 25505484